CLINICAL TRIAL: NCT06609057
Title: Cooking for Your Health in Southern New Mexico
Brief Title: Cooking for Your Health in Southern New Mexico: an 8-week, Bilingual (English and Spanish) Nutritional Intervention in Adults Living in Doña Ana and Otero Counties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New Mexico State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1124544; NCI-2024-06525 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20558 (Other: Fred Hutch/University of Washington Cancer Consortium); U54CA132381 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dietary Carcinogenesis; Nutrition, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (nutrition intervention) (Experimental): Participants attend Cooking for Your Health in Southern New Mexico intervention sessions, consisting of 15-30 minutes of pre-work (watching an educational video and/or practicing a new culinary skill), 60 minutes of hands-on experiential cooking and culinary session in a teaching kitchen, and a 60 minute meal that includes group discussion of educational information, QW for 6 weeks.
  Interventions: Other: Nutritional Intervention; Other: Questionnaire Administration; Other: Survey Administration; Other: Discussion

INTERVENTIONS:
Other: Nutritional Intervention — Receive Cooking for Your Health in Southern New Mexico intervention
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Discussion — Ancillary studies
  Other Names: Discuss

SUMMARY:
This clinical trial evaluates a nutritional intervention called Cooking for Your Health in Southern New Mexico for improving diet quality and knowledge related to nutrition and cancer prevention among individuals living in the Southern region of New Mexico. New Mexico border communities have high rates of cancer and obesity, both exacerbated by poor diet quality. Traditional Mexican diets are high in fruit, vegetables, and fiber, but are intensive to prepare and not practical for many families living in New Mexico now. Vegetable oils, such as canola, safflower, and sunflower oils, are commonly used in cooking within the regional New Mexican community because they are inexpensive and readily available; however, they may not be as healthy as other options. Interventions focused on teaching proper cooking techniques and raising awareness about nutritious foods have shown positive behavior changes, including greater preference for healthier foods, increased confidence in food preparation and cooking a balanced meal, and higher vegetable variety and availability in the home. This study may help identify effective and culturally relevant real-world strategies to improve knowledge, skills, behaviors, and access to resources to improve nutrient intake, with the long-term goal of decreasing cancer risk and chronic disease risk in southern New Mexican communities.

DETAILED DESCRIPTION:
OUTLINE:

Participants attend Cooking for Your Health in Southern New Mexico intervention sessions, consisting of 15-30 minutes of pre-work (watching an educational video and/or practicing a new culinary skill), 60 minutes of hands-on experiential cooking and culinary session in a teaching kitchen, and a 60 minute meal that includes group discussion of educational information, once a week (QW) for 6 weeks.

After completion of study intervention, participants are followed up at week 8 and 10.

The study originally closed to accrual in May 2025, with 33 participants enrolled. Following a modification to add a second cohort, the study reopened to accrual in October 2025.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Part I: Fluent in English (Otero and Doña Ana Counties); Part II: Fluent in English (Otero County) and fluent in Spanish (Doña Ana County)
* Able to understand and willing to sign a written informed consent in either English or in Spanish (Part II only: Doña Ana County only)
* Access to phone for study contacts
* Be willing and able to attend the 6 in-person classes
* Access to internet to complete study assessments and access study website
* Willingness to participate in all study activities
* Completion of all baseline data collection activities
* No prior clinical diagnosis of diabetes

Exclusion Criteria:

* Under 18 years of age, or over 70 years of age
* Not fluent in either Spanish or English (Part II only: Doña Ana County only)
* Unable to understand or unwilling to sign written informed consents in English or in Spanish (Part II only: Doña Ana County only)
* No access to phone
* Unwilling or unable to attend the 6 in person classes
* No access to internet
* Unwilling to participate in all study activities
* Unable to complete all run in activities
* Prior clinical diagnosis of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Accrual rate | Within 6 months of trial activation
  The intervention will be considered feasible if accrual goals are met within 6 months of trial activation. Will be summarized using descriptive statistics. Results will be assessed separately for Part I and Part II, as well as for both groups combined.
Engagement | Up to 8 weeks
  The intervention will be considered feasible if >= 70% of participants attend >= 70% of sessions. Will be summarized using descriptive statistics. Results will be assessed separately for Part I and Part II, as well as for both groups combined.
Retention | At week 8
  The intervention will be considered feasible if >= 70% of participants complete the week 8 food frequency questionnaire. Will be summarized using descriptive statistics. Results will be assessed separately for Part I and Part II, as well as for both groups combined.
Acceptability | Up to 8 weeks
  The intervention will be considered feasible if >= 70% or more of participants state that the program and study processes were acceptable, appropriate, and feasible. Acceptability will assess: intervention pre-work and in-class work activities, as well as specific data collection methods. Will be summarized using descriptive statistics. Results will be assessed separately for Part I and Part II, as well as for both groups combined.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, ND, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- New Mexico State University, Las Cruces, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT06609057/ICF_000.pdf